CLINICAL TRIAL: NCT00734591
Title: An Observational Follow-Up Study Of Patients Previously Enrolled In Exubera Controlled Clinical Trials
Brief Title: Follow-Up Study for Exubera
Acronym: FUSE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A2171121
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Results first posted 2012-10-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes Mellitus
Keywords: Observational Study Exubera
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exubera

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Previously treated with Exubera
  Interventions: Drug: Exubera
- Previously treated with comparator: Subjects who had been treated with a comparator (other diabetes treatment such as injected insulin) in a prior Exubera controlled trial.
  Interventions: Other: Randomized diabetes therapy

INTERVENTIONS:
Drug: Exubera — Subjects who had been treated with Exubera in a prior Exubera controlled trial. Following initial use of randomized treatment, physicians and subjects were free to change regimens and dosing based on subject response to assigned treatment (as consistent with routine practice).
  Groups: Previously treated with Exubera
Other: Randomized diabetes therapy — Subjects who had been treated with a comparator (other diabetes treatment including one or more of: subcutaneous insulin, sulfonylureas, biguanides, or thiazolinediones) in a prior Exubera controlled trial.
  Following initial use of randomized treatment, physicians and subjects were free to change regimens and dosing based on subject response to assigned treatment (as consistent with routine practice).
  Groups: Previously treated with comparator

SUMMARY:
In studies of Exubera in persons with diabetes, lung cancer occurred in a few more people who were taking Exubera than in people who were taking other diabetes medicines. All subjects diagnosed with lung cancer had a history of smoking and the number of lung cancer cases observed fell within the expected range based on population-based data. There is currently not enough information to determine if any of the observed lung cancer cases were related to Exubera use, therefore, the study is being conducted to further investigate whether Exubera use makes the appearance of lung cancer more likely.

DETAILED DESCRIPTION:
Both retrospective and prospective components All subjects who participated in one of the 17 included Exubera clinical trials will be invited to participate in the current study.

ELIGIBILITY:
Inclusion Criteria:

* Previously participated in an eligible Exubera clinical trial
* Willing to provide study doctor with at least one alternate contact person

Exclusion Criteria:

* Participated in an investigational study of an unapproved drug since completing the Exubera trial
* Ever used an other (non-Exubera) inhaled insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who participated in a controlled trial of Exubera active within the last five years (17 protocols total)
Sampling Method: Non-Probability Sample
Enrollment: 7439 (Actual)
Dates: Start 2008-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (284):
- United States (114):
  - Pfizer Investigational Site, Bay Minette, Alabama
  - Pfizer Investigational Site, Graysville, Alabama
  - Pfizer Investigational Site, Pell City, Alabama
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Forrest City, Arkansas
  - Pfizer Investigational Site, Berkeley, California
  - Pfizer Investigational Site, Concord, California
  - Pfizer Investigational Site, El Cajon, California
  - Pfizer Investigational Site, Encino, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Fullerton, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Rolling Hills Estates, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Jose, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Santa Barbara, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Golden, Colorado
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, Milford, Connecticut
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Chiefland, Florida
  - Pfizer Investigational Site, Green Cove Springs, Florida
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Lake City, Florida
  - Pfizer Investigational Site, Lake Mary, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Opa-locka, Florida
  - Pfizer Investigational Site, Saint Cloud, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Conyers, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Hayden Lake, Idaho
  - Pfizer Investigational Site, Greenville, Illinois
  - Pfizer Investigational Site, Normal, Illinois
  - Pfizer Investigational Site, Olympia Fields, Illinois
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Fishers, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Mount Sterling, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Elkton, Maryland
  - Pfizer Investigational Site, Glen Burnie, Maryland
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Clinton, Michigan
  - Pfizer Investigational Site, Flint, Michigan
  - Pfizer Investigational Site, Muskegon, Michigan
  - Pfizer Investigational Site, Saint Cloud, Minnesota
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Incline Village, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Belvidere, New Jersey
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Babylon, New York
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Minneola, New York
  - Pfizer Investigational Site, New Hartford, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Asheboro, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Morehead City, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Tabor City, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Marietta, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Fogelsville, Pennsylvania
  - Pfizer Investigational Site, Hanover, Pennsylvania
  - Pfizer Investigational Site, Harrisburg, Pennsylvania
  - Pfizer Investigational Site, Jeannette, Pennsylvania
  - Pfizer Investigational Site, Jersey Shore, Pennsylvania
  - Pfizer Investigational Site, Lansdale, Pennsylvania
  - Pfizer Investigational Site, Melrose Park, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, North Myrtle Beach, South Carolina
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Kaufman, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, San Marcos, Texas
  - Pfizer Investigational Site, Stephenville, Texas
  - Pfizer Investigational Site, Webster, Texas
  - Pfizer Investigational Site, South Burlington, Vermont
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Federal Way, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Burnsville, West Virginia
- Argentina (2):
  - Pfizer Investigational Site, Capital Federal, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires
- Australia (5):
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Wollongong, New South Wales
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Box Hill, Victoria
  - Pfizer Investigational Site, Melbourne, Victoria
- Pfizer Investigational Site, Vienna, Austria
- Belgium (6):
  - Pfizer Investigational Site, Bornem
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Liège
- Brazil (3):
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (22):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Corunna, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Oakville, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Smiths Falls, Ontario
  - Pfizer Investigational Site, Thornhill, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Gatineau, Quebec
  - Pfizer Investigational Site, Greenfield Park, Quebec
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Trois-Rivières, Quebec
- Pfizer Investigational Site, Zagreb, Croatia
- Denmark (3):
  - Pfizer Investigational Site, Aarhus
  - Pfizer Investigational Site, Copenhagen
  - Pfizer Investigational Site, Herning
- Estonia (3):
  - Pfizer Investigational Site, Viljandi, Viljandi Mk.
  - Pfizer Investigational Site, Pärnu
  - Pfizer Investigational Site, Tallinn
- Finland (4):
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Lahti
  - Pfizer Investigational Site, Lohja
  - Pfizer Investigational Site, Oulu
- France (10):
  - Pfizer Investigational Site, Corbeil-Essonnes, France
  - Pfizer Investigational Site, Amiens
  - Pfizer Investigational Site, Armentières
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Bondy
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Chartres
  - Pfizer Investigational Site, Lorient
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Rennes
- Germany (36):
  - Pfizer Investigational Site, Altenburg
  - Pfizer Investigational Site, Aschaffenburg
  - Pfizer Investigational Site, Bad Doberan
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Chemnitz
  - Pfizer Investigational Site, Datteln
  - Pfizer Investigational Site, Dortmund
  - Pfizer Investigational Site, Eisenach
  - Pfizer Investigational Site, Emden
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Falkensee
  - Pfizer Investigational Site, Friedberg
  - Pfizer Investigational Site, Fulda
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hohenmölsen
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Leverkusen
  - Pfizer Investigational Site, Marl
  - Pfizer Investigational Site, Meissen
  - Pfizer Investigational Site, Mittweida
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Neuss
  - Pfizer Investigational Site, Reinfeld
  - Pfizer Investigational Site, Riesa
  - Pfizer Investigational Site, Rossach
  - Pfizer Investigational Site, Schlüchtern
  - Pfizer Investigational Site, Siegen
  - Pfizer Investigational Site, Suhl
  - Pfizer Investigational Site, Surwold
  - Pfizer Investigational Site, Villingen-Schwenningen
  - Pfizer Investigational Site, Wangen
  - Pfizer Investigational Site, Wangen / Allgaeu
  - Pfizer Investigational Site, Warburg
  - Pfizer Investigational Site, Wiesbaden
- Greece (2):
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Thessaloniki
- Italy (8):
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Udine
- Mexico (2):
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Monterrey, Nuevo León
- Netherlands (5):
  - Pfizer Investigational Site, 's-Hertogenbosch
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Beek
  - Pfizer Investigational Site, Eindhoven
  - Pfizer Investigational Site, Venlo
- Norway (4):
  - Pfizer Investigational Site, Fornebu
  - Pfizer Investigational Site, Hønefoss
  - Pfizer Investigational Site, Skedsmokorset
  - Pfizer Investigational Site, Stavanger
- Poland (4):
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Łask
- Portugal (4):
  - Pfizer Investigational Site, Aveiro
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
  - Pfizer Investigational Site, Torres Vedras
- Slovakia (3):
  - Pfizer Investigational Site, Banská Bystrica
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Martin
- South Africa (2):
  - Pfizer Investigational Site, Houghton Estate, Gauteng
  - Pfizer Investigational Site, Umhlanga, KwaZulu-Natal
- Spain (12):
  - Pfizer Investigational Site, Santiago de Compostela, A Coruña
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Granada, Granada
  - Pfizer Investigational Site, Las Palmas, Las Palmas de Gran Canaria
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Alzira, Valencia
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Bilbao, Vizcaya
- Sweden (9):
  - Pfizer Investigational Site, Borås
  - Pfizer Investigational Site, Forshaga
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Härnösand
  - Pfizer Investigational Site, Helsingborg
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Vaxjo
- United Kingdom (19):
  - Pfizer Investigational Site, Penzance, Cornwall
  - Pfizer Investigational Site, St Austell, Cornwall
  - Pfizer Investigational Site, Plymouth, Devon
  - Pfizer Investigational Site, Letchworth Garden City, Hertfordshire
  - Pfizer Investigational Site, Ashford, Middlesex
  - Pfizer Investigational Site, Headington, Oxford
  - Pfizer Investigational Site, Weybridge, Surrey
  - Pfizer Investigational Site, Woking, Surrey
  - Pfizer Investigational Site, Rugby, Warwickshire
  - Pfizer Investigational Site, Warminster, Wiltshire
  - Pfizer Investigational Site, Sheffield, Yorkshire
  - Pfizer Investigational Site, Bath
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Bolton
  - Pfizer Investigational Site, Canterbury
  - Pfizer Investigational Site, Leicester
  - Pfizer Investigational Site, Newcastle upon Tyne
  - Pfizer Investigational Site, Salford
  - Pfizer Investigational Site, Westbury

REFERENCES:
- [Derived] Gatto NM, Koralek DO, Bracken MB, Duggan WT, Lem J, Klioze S, Koch GG, Wise RA, Cohen RB, Jackson NC. Lung Cancer-Related Mortality With Inhaled Insulin or a Comparator: Follow-Up Study of patients previously enrolled in Exubera Controlled Clinical Trials (FUSE) Final Results. Diabetes Care. 2019 Sep;42(9):1708-1715. doi: 10.2337/dc18-2529. Epub 2019 Jul 22. PMID 31331907
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171121&StudyName=Follow-Up%20Study%20for%20Exubera

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had retrospective and prospective components. Individuals who participated in Exubera-controlled trials that were still active in 2003 or later participated in the retrospective part of this study (Follow-Up Study for Exubera; FUSE). Individuals from sites participating in the prospective part of FUSE were eligible.
Groups:
- Previously Randomized to Exubera: Participants randomized to Exubera® (inhalable form of recombinant human [rh] insulin) per protocol in a prior Exubera-controlled clinical trial. There was no active study medication used in FUSE. During prospective follow-up all participants received treatment for diabetes mellitus per routine clinical practice.
- Previously Randomized to Comparator: Participants randomized to comparator (Type 1 or Type 2 diabetes mellitus treatments such as injected insulin or oral agent therapy) in a prior Exubera-controlled trial. There was no active study medication used in FUSE. During prospective follow-up all participants received treatment for diabetes mellitus per routine clinical practice.
Period: Retrospective Period
Arm/Group | Previously Randomized to Exubera | Previously Randomized to Comparator
Started | 3875 | 3564
Completed | 3875 | 3564
Not Completed | 0 | 0
Period: Screening for Prospective Period
Arm/Group | Previously Randomized to Exubera | Previously Randomized to Comparator
Started | 3875 | 3564
Completed | 1358 | 1273
Not Completed | 2517 | 2291
Not completed — Site did not participate | 1604 | 1488
Not completed — Patient at partic. site not enrolled | 913 | 803
Period: Prospective Period
Arm/Group | Previously Randomized to Exubera | Previously Randomized to Comparator
Started | 1358 | 1273
Completed | 1307 | 1229
Not Completed | 51 | 44
Not completed — Withdrawal by Subject | 11 | 9
Not completed — Lost to Follow-up | 37 | 33
Not completed — Study Terminated | 1 | 0
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Previously Randomized to Exubera | Previously Randomized to Comparator | Total
Number analyzed (Participants) | 3875 | 3564 | 7439
Age Continuous [Mean (Standard Deviation); unit: years] — Mean age at original trial
  years | 54.8 (12.1) | 54.7 (12.6) | 54.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1677 | 1557 | 3234
  Male | 2198 | 2007 | 4205
Smoking status [Number; unit: participants] — Reported as number of participants who never smoked (never-smoker) and those who have ever smoked (ever-smoker) includes former smokers and current smokers.
  participants
    Never-smoker | 2194 | 2031 | 4225
    Ever-smoker | 1681 | 1533 | 3214

OUTCOME MEASURES:

1. Primary Outcome: Rate of Primary Lung Cancer Mortality
Description: Reported deaths from primary lung cancer were adjudicated and classified into 4 categories: highly likely (clinical, radiographic, and/or histological data consistent with primary lung cancer); likely (some information may have been missing for definite diagnosis); unlikely; insufficient information. Highly likely and likely cases used to report rate and rate ratio of primary lung cancer mortality. Includes events from the start of the original trial to the end of FUSE.
Time Frame: Baseline from original trial up to Year 2 of this study
Population: Entire study population: all randomized participants (retrospective).
Measure: Number (95% Confidence Interval); unit: Deaths per 1000 patient years (PY)
Arm/Group | Previously Randomized to Exubera | Previously Randomized to Comparator
Number analyzed (Participants) | 3875 | 3654
Deaths per 1000 patient years (PY) | 0.48 [0.17 to 1.04] | 0.17 [0.02 to 0.61]
Statistical Analysis 1: Comparison: Previously Randomized to Exubera vs Previously Randomized to Comparator; Test type: Superiority or Other; Exact method = 2.81, 95% CI 2-sided [0.50 to 28.46] — Incidence density ratio confidence interval derived from exact methods utilizing exact binomial limits and ratio of exposures

2. Secondary Outcome: Rate of Primary Lung Cancer Mortality Among Former Smokers
Description: as for outcome 1
Time Frame: Baseline from original trial up to Year 2 of this study
Population: Subset of the entire study population who were former smokers.
Measure: Number (95% Confidence Interval); unit: Deaths per 1000 PY
Arm/Group | Previously Randomized to Exubera | Previously Randomized to Comparator
Number analyzed (Participants) | 1681 | 1533
Deaths per 1000 PY | 0.94 [0.30 to 2.18] | 0.41 [0.05 to 1.48]
Statistical Analysis 1: Comparison: Previously Randomized to Exubera vs Previously Randomized to Comparator; Test type: Superiority or Other; Exact method = 2.29, 95% CI 2-sided [0.37 to 24.01] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Rate of All-cause Mortality
Description: The rate and rate ratio of all-cause mortality that occurred anytime from the start of the original trial to the end of FUSE.
Time Frame: Baseline from original trial up to Year 2 of this study
Population: Entire study population
Measure: Number (95% Confidence Interval); unit: Deaths per 1000 PY
Arm/Group | Previously Randomized to Exubera | Previously Randomized to Comparator
Number analyzed (Participants) | 3875 | 3564
Deaths per 1000 PY | 6.03 [4.75 to 7.55] | 7.37 [5.90 to 9.09]
Statistical Analysis 1: Comparison: Previously Randomized to Exubera vs Previously Randomized to Comparator; Test type: Superiority or Other; Cox Proportional Hazard = 0.81, 95% CI 2-sided [0.60 to 1.10]

4. Secondary Outcome: Rate of Primary Lung Cancer Diagnosis
Description: The rate and rate ratio of lung cancer adjudicated as highly likely (clinical, radiographic, and/or histological data consistent with primary lung cancer) or likely (some information may have been missing for definite diagnosis) to be newly diagnosed primary lung cancer that occurred anytime from the start of the original trial to the end of FUSE.
Time Frame: Baseline from original trial up to Year 2 of this study
Population: Entire study population
Measure: Number (95% Confidence Interval); unit: Lung Cancer per 1000 PY
Arm/Group | Previously Randomized to Exubera | Previously Randomized to Comparator
Number analyzed (Participants) | 3875 | 3564
Lung Cancer per 1000 PY | 1.07 [0.55 to 1.87] | 0.29 [0.06 to 0.84]
Statistical Analysis 1: Comparison: Previously Randomized to Exubera vs Previously Randomized to Comparator; Test type: Superiority or Other; Exact method = 3.75, 95% CI 2-sided [1.01 to 20.68] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: Adverse events were not collected.
Arm/Group | Previously Randomized to Exubera | Previously Randomized to Comparator
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Detection and/or reporting bias possible in continuous analysis (presented here) of lung cancer mortality and lung cancer incidence endpoints. Study had insufficient power to draw clear statistical conclusions due to small number of events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.